CLINICAL TRIAL: NCT06443866
Title: CLINICAL UTILITY AND FEASIBILITY OF I-124 PET/CT IMAGING AND DOSIMETRY IN PATIENTS WITH THYROID CANCER
Brief Title: I-124 PET/CT Imaging and Dosimetry for RAI-Naïve or Refractory Thyroid Cancer
Status: Recruiting | Type: Observational
Sponsor: Miami Cancer Research Center, Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: MTOCP03; MBK funding (Other: MiamiCancerRC)
Record Dates: First submitted 2024-05-23; First posted 2024-06-05 (Actual); Last update posted 2024-06-05 (Actual); Status verified 2024-05

CONDITIONS: Thyroid Cancer; RAI-Refractory Thyroid Cancer
Keywords: Thyroid Cancer; RAI-Refractory Thyroid Cancer; Redifferentiation Therapy
MeSH Terms: conditions — Thyroid Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

GROUPS / COHORTS (1):
- Thyroid Cancer patients, RAI-naive or refractory
  Interventions: Diagnostic Test: Disease status detection; Diagnostic Test: Theranostic dosimetry; Drug: I-124 PET/CT imaging

INTERVENTIONS:
Diagnostic Test: Disease status detection — RAI dose determination
Diagnostic Test: Theranostic dosimetry — Theranostic dosimetric evaluation for optimization of RAI therapy of thyroid cancer
Drug: I-124 PET/CT imaging — Theranostic dosimetry for optimization of RAI therapy for Thyroid Cancer

SUMMARY:
The objective of this study is to demonstrate the clinical utility of I-124 PET/CT imaging and dosimetry in patients with thyroid cancer including 1) Evaluation of extent (volume and pattern) of remnant tissue in post total thyroidectomy setting and distinction of nodal metastases vs remnant tissue for determination of indication for RAI ablation, 2) Evaluation of response to RAI remnant ablation, 3) Evaluation for suspected occult recurrent/metastatic disease, 4) Evaluation of extent of disease in patients with known metastatic disease and 5) Evaluation of RAI avidity of recurrent/metastatic thyroid cancer and response to treatment with thyroid kinase inhibitors (TKI).

Patients who underwent total thyroidectomy for thyroid cancers are studied. Patients who are newly diagnosed, as well as those who have known or suspected to have recurrent or metastatic disease are eligible. Patients receiving TKI treatment are eligible for evaluation prior to and after the treatment. The patients who are considered for TKI/MAPK treatments undergo pre and post treatment with clinically determined oncoprotein/TKR therapeutic agent(s), including multi-TKI, selective BRAF, MEK, PI3K or ERK inhibitors or combination treatments.

ELIGIBILITY:
Inclusion Criteria

* Post-total thyroidectomy patients with diagnosis of thyroid cancer, any histology, subtype, any ATA risk category, for evaluation for residual disease, cervical or remote metastatic disease
* Patients with known or suspected recurrent/metastatic thyroid cancer, identified by ultrasound (US), CT/MR/FDG-PET|CT or elevated thyroglobulin (Tg).
* Pretreatment and post-treatment evaluation of patients with thyroid cancer deemed RAI-indifferent/refractory who are considered for TKI
* Age ≥ 18
* Ability and willingness to give a written consent
* Life expectancy > 3 months
* ECOG performance status ≤ 2

Exclusion Criteria

* Cancers metastatic to thyroid
* Age < 18
* Inability or unwillingness to give a written consent
* Life expectancy < 3 months
* ECOG performance status ≥ 3
* Pregnant and nursing women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (18 and older) with thyroid cancer
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2029-01-31 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Identification and characterization of RAI uptake pattern and kinetics | 5 years
  Measurements:
  1. Administered activity
  2. Cumulated activity
  3. Standard uptake value
  Calculations:
  1. Radiation absorbed dose to the target
  Correlations to be reported:
  1. Administered activity vs absorbed dose
  2. Absorbed dose vs response
  3. SUV at 48h vs response

CONTACTS AND LOCATIONS:
Overall Officials: Seza Gulec, MD, Principal Investigator — CEO, MCRC
Locations (1):
- Miami Cancer Research Center, North Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No